CLINICAL TRIAL: NCT03575273
Title: The Impact of Methadone Maintenance Therapy on Food Intake and Food Reward Processing in Opioid Dependence: An Event-related Brain Potential Study
Brief Title: The Impact of Methadone Maintenance Therapy on Food Reward Processing in Opioid Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Mid-Atlantic Nutrition Obesity Research Center (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00092798; P30DK072488 (NIH)
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Opioid Dependence; Obesity
Keywords: methadone; opioid dependence; obesity; food reward; olfactory
MeSH Terms: conditions — Opioid-Related Disorders; Obesity; Anosmia | interventions — potassium channel subfamily K member 3; Hunger

STUDY DESIGN:
Intervention Model Description: The investigators will recruit thirty individuals meeting criteria for opioid dependence of which 15 will be receiving MMT (O+MMT) and 15 will be on no opioid agonist therapy (O-MMT). The investigators will attempt to match the O-MMT group to the O+MMT group for clinical characteristics and smoking burden. Fifteen obese/overweight adults without history of opioid/substance use will be matched to the patient groups for age, gender, education, smoking and BMI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Opioid dependence receiving methadone (Experimental): Patients with a history of opioid dependence receiving methadone maintenance therapy will be administered Sniffin' Sticks Odor Identification and Hedonic Scale, Sucrose Taste Preference Assessment, Food Preferences Task, Progressive Ratio Task, Clinical Electrophysiology, and Standardized Meal and Hunger and Satiety Ratings
  Interventions: Behavioral: Sniffin' Sticks Odor Identification and Hedonic Scale; Behavioral: Sucrose Taste Preference Assessment; Behavioral: Food Preferences Task; Behavioral: Progressive Ratio (PR) Task; Procedure: Clinical Electrophysiology; Dietary Supplement: Standardized Meal and Hunger and Satiety Ratings
- Opioid dependence not on methadone (Experimental): Patients with a history of opioid dependence not current receiving methadone maintenance therapy will be administered Sniffin' Sticks Odor Identification and Hedonic Scale, Sucrose Taste Preference Assessment, Food Preferences Task, Progressive Ratio Task, Clinical Electrophysiology, and Standardized Meal and Hunger and Satiety Ratings
  Interventions: Behavioral: Sniffin' Sticks Odor Identification and Hedonic Scale; Behavioral: Sucrose Taste Preference Assessment; Behavioral: Food Preferences Task; Behavioral: Progressive Ratio (PR) Task; Procedure: Clinical Electrophysiology; Dietary Supplement: Standardized Meal and Hunger and Satiety Ratings
- Healthy controls (Active Comparator): Healthy controls without history of opioid use will be administered Sniffin' Sticks Odor Identification and Hedonic Scale, Sucrose Taste Preference Assessment, Food Preferences Task, Progressive Ratio Task, Clinical Electrophysiology, and Standardized Meal and Hunger and Satiety Ratings
  Interventions: Behavioral: Sniffin' Sticks Odor Identification and Hedonic Scale; Behavioral: Sucrose Taste Preference Assessment; Behavioral: Food Preferences Task; Behavioral: Progressive Ratio (PR) Task; Procedure: Clinical Electrophysiology; Dietary Supplement: Standardized Meal and Hunger and Satiety Ratings

INTERVENTIONS:
Behavioral: Sniffin' Sticks Odor Identification and Hedonic Scale — This task measures odor identification accuracy and perceived pleasantness of odors.
Behavioral: Sucrose Taste Preference Assessment — This task measures participant ratings of sucrose preference.
Behavioral: Food Preferences Task — Participants rate images of various food stimuli. Variables derived include relative preferences and reaction time (in milliseconds).
Behavioral: Progressive Ratio (PR) Task — In the PR task, the subject is required to make an increasing number of operant responses for each successive reward
Procedure: Clinical Electrophysiology — To examine motivated attention in response to food stimuli, brain electrophysiology via event related potentials (ERPs) will be assessed while participants view and rate images of food and non-food items.
Dietary Supplement: Standardized Meal and Hunger and Satiety Ratings — Participants will receive a standardized meal and complete hunger and satiety ratings.

SUMMARY:
Methadone maintenance therapy (MMT) has shown clear efficacy for relieving opioid withdrawal symptoms and reducing the morbidity and mortality of opioid dependence. A notable phenomenon associated with MMT is increased food intake, enhanced sweet preferences, and weight gain. The underlying neural mechanisms for opioid-related overconsumption are not well understood but are thought to arise from role in 1) increasing the palatability and hedonic aspects of food and 2) diminishing satiety signaling systems. In the proposed project, the investigators will examine methadone's potential role in opioid-related overconsumption of food. The investigators propose to examine eating behavior, sucrose preferences, and an event-related potential (ERP) component that is induced by appetitive motivation for highly rewarding foods in patients with a history of opioid dependence receiving methadone maintenance therapy (O+MMT) and not receiving opioid agonist therapy (O-MMT). A matched sample of obese and overweight adults without history of opioid use (HOC) will also be examined.

DETAILED DESCRIPTION:
Methadone maintenance therapy (MMT) has shown clear efficacy for relieving opioid withdrawal symptoms and reducing the morbidity and mortality of opioid dependence. A notable phenomenon associated with MMT is increased food intake, enhanced sweet preferences, and weight gain. The underlying neural mechanisms for opioid-related overconsumption are not well understood but are thought to arise from role in 1) increasing the palatability and hedonic aspects of food and 2) diminishing satiety signaling systems. In the proposed project, the investigators will examine methadone's potential role in opioid-related overconsumption of food. The investigators propose to examine eating behavior, sucrose preferences, and an event-related potential (ERP) component that is induced by appetitive motivation for highly rewarding foods in patients with a history of opioid dependence receiving methadone maintenance therapy (O+MMT) and not receiving opioid agonist therapy (O-MMT). A matched sample of obese and overweight adults without history of opioid use (HOC) will also be examined. Specifically, group differences in food intake and eating behaviors in the O+MMT group relative to individuals in the O-MMT and HOC group will be examined. Individuals will complete 24-hour dietary food recalls and inventories to characterize eating behavior and food addiction. Participants will complete psychophysical measures of chemosensory functioning of sucrose preference and pleasantness and identification ratings for odors varying in participants' hedonic characteristics. Individuals will also complete validated computer tasks to assess food preferences. Differences in cortical ERPs for high-reward food relative to low-reward food and non-food items will be examined. Event-related potentials will be recorded as participants view photos of rewarding and non-rewarding food items, as well as non-food items. ERP components that index sustained attentional engagement will be measured and compared.

ELIGIBILITY:
Inclusion criteria:

* English-speaking individuals
* Must be between 18 and 60 years of age
* For the O+MMT group, participants must be receiving MMT for at least 3 months
* For the O-MMT group, participants must have concluded their MMT (if applicable) at least three months prior to the date of the screening visit.

Exclusion criteria:

* Individuals may not have a history of major neurological disorders
* No unstable medical issues that would affect appetite or blood glucose
* No pervasive developmental disorder or intellectual disability
* No significant visual/auditory impairment
* No history or current episode of psychosis
* No current opioid abuse
* No current antipsychotic medication use
* No major conditions that affect chemosensory function (e.g., history of nasal fracture or respiratory infection)
* Individuals with contraindication for the EEG will be excluded
* Individuals who are current pregnant or breastfeeding will not be enrolled
* For HOC, individuals with history of opioid dependence or current or past psychiatric disorders will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Event-related potentials measured via BrainVision actiCHamp system | At baseline visit
  Cortical ERPs for high-reward food relative to low-reward food and non-food items will be measured using a BrainVision actiCHamp system (32-channel amplifier). For each group, the grand averages and standard deviations for the late positive potential will be calculated. Group differences in LPP will be assessed within and between picture categories for each arm of the study.

SECONDARY OUTCOMES:
Chemosensory Processing | At baseline visit
  For the odorants, participants provide a rating of intensity and pleasantness based on a -5 to 5 point scale for each of the 16 markers. Afterwards, averages of all 16 marker scores will be calculated for the mean ratings of intensity and pleasantness. Odor identification accuracy will be assessed for each marker, with the score representing the total items correct out of 16.
Food Preferences Task | At baseline visit
  Participants are showed images of high fat savory, low fat savory, high fat sweet, and low fat sweet foods. Participants must select one of the two pictures to answer the question "which food item do you most want to eat right now." Selection averages of each category and time for selection, for each arm of the study, are automatically calculated by E-Prime software.
Progressive Ratio Task | At baseline visit
  Participants begin with 20 M&Ms and a computer prompt that specifies how many times the mouse must be clicked to earn a piece of candy. Participants can earn as little as desired. The click ratio starts at 10 and geometrically increases in increments of 2 (i.e., 10, 20, 40, 80, etc.). The computer program E-Prime automatically records the participant's work capacity and the administrator records the number of M&Ms left in the cup.

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Kamath, Ph.D., Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Broadway Center for Addictions, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No